CLINICAL TRIAL: NCT04659278
Title: A Post Marketing Study to Evaluate the Safety and Efficacy of Endourage Complete Spectrum Oral Mucosal Drops (OMD) in Adults Desiring a Reduction in Ethanol Use
Brief Title: Endourage Complete Spectrum Oral Mucosal Drops (OMD) in Adults Desiring a Reduction in Ethanol Use
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study has been placed on hold
Sponsor: Endourage, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CSP ENDO 401-2020
Record Dates: First submitted 2020-10-03; First posted 2020-12-09 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Drinking; Alcohol Use, Unspecified; Alcohol Abstinence; Alcohol-Related Disorders
MeSH Terms: conditions — Alcohol Drinking; Alcohol Abstinence; Alcohol-Related Disorders | interventions — peppermint oil

STUDY DESIGN:
Intervention Model Description: This is a 112-day, double-blind, placebo-controlled clinical trial evaluating the safety and efficacy of Endourage 1200 mg Complete Spectrum Oral Mucosal Drops (OMD ™). A total of 32 study participants will be enrolled.
  Placebo (Hemp seed oil and peppermint flavoring)
  Isolate (CBD no terpenes Hemp seed oil [slightly lower concentration of CBD ratio])
  Endourage OMD (Full flower extract with a 1:1 ratio of cannabis terpenes, Hemp seed oil and peppermint flavoring)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be double-blind; neither the Investigator nor the study participant will know to which study treatment arm the participant is assigned. All 3 study treatments will be packaged in identical bottles and similar labelling. Study treatment dispensing and return will be managed centrally; study treatment will be mailed directly to study participants. The 2 control test articles have been designed and flavored to look and taste like OMD study product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 Placebo (Placebo Comparator): Placebo Isolate Placebo (Hemp seed oil and peppermint flavoring)
  Interventions: Dietary Supplement: Isolate; Other: Placebo; Dietary Supplement: Peppermint Oil, masking flavor
- Group 2 Isolate Comparator (Active Comparator): Isolate Placebo Isolate (CBD no terpenes Hemp seed oil [slightly lower concentration of CBD ratio])
  Interventions: Dietary Supplement: Isolate; Other: Placebo; Dietary Supplement: Peppermint Oil, masking flavor
- Group 3 Placebo Comparator (Placebo Comparator): Placebo OMD Endourage OMD (Full flower extract with a 1:1 ratio of cannabis terpenes, Hemp seed oil and peppermint flavoring)
  Interventions: Dietary Supplement: Endourage 1200 mg OMD ™ Oral Mucosal Drops; Other: Placebo; Dietary Supplement: Peppermint Oil, masking flavor
- Group 4 Experimental Placebo (Experimental): OMD Placebo Endourage OMD (Full flower extract with a 1:1 ratio of cannabis terpenes, Hemp seed oil and peppermint flavoring)
  Interventions: Dietary Supplement: Endourage 1200 mg OMD ™ Oral Mucosal Drops; Other: Placebo; Dietary Supplement: Peppermint Oil, masking flavor

INTERVENTIONS:
Dietary Supplement: Endourage 1200 mg OMD ™ Oral Mucosal Drops — The CBD/THC ratio of OMD 1200 is 14:1 and the CBD/Terpene ratio is 1:1. Each ¼ dropper contains 10.2 mg of CBD and 0.7 mg of THC. The total % THC is 0.28%. These ratios indicate that the product will not cause euphoria.
  Other Names: OMD-1200; OMD 1200; Endourage OMD 1200
  Arms: Group 3 Placebo Comparator; Group 4 Experimental Placebo
Dietary Supplement: Isolate — The isolate formulation contains 0% cannabinoids (CBD 0.00%; CBDa 0.00%; detla 9 THC 0.00%; THCa 0.00%).
  Arms: Group 1 Placebo; Group 2 Isolate Comparator
Other: Placebo — Total CBD = CBD + (CBD-A * 0.877). Total THC = THCA-A * 0.877 + Delta 9 THC, ND = <LOQ, T-Caryophyllene = Trans-Caryophyllene, <LOQ = Less Than Limit of Quantitation, QNS = Quantity Not Sufficient. (%) = Percent, (ppm) = Parts per Million, (ppb) = Parts per Billion, (μg/Kg) = Microgram per Kilogram, (mg/g) = Milligram per Gram, ppm = (μg/g), ppb = (μg/kg),
Dietary Supplement: Peppermint Oil, masking flavor — Mentha piperita Leaf /Stem Oil; Physical state: Liquid. Color: Colorless to pale yellow; Characteristic peppermint odor; Not dangerous goods.
  Other Names: Peppermint Oil; Peppermint Oil, Natural

SUMMARY:
This is the first clinical trial of Endourage OMD 1200 for persons desiring to reduce their alcohol consumption.

DETAILED DESCRIPTION:
CBD is the second most abundant component of the cannabis plant after tetrahydrocannabinol (THC). Unlike THC, CBD does not get users high, but there is some evidence suggesting that it might have anti-anxiety, anticonvulsant, anti-inflammatory and immune boosting, antioxidant effects.

Currently, the only CBD product approved by the Food and Drug Administration is a prescription oil called Epidiolex (Greenwich Biosciences, Inc. 2018). It is approved to treat two types of epilepsy. Aside from Epidiolex, state laws on the use of CBD vary. While CBD is being studied as a treatment for a wide range of conditions, including Parkinson's disease, schizophrenia, diabetes, multiple sclerosis and anxiety, and addiction, research supporting the drug's benefits is still limited.

CBD use carries some risks. Though it is often well-tolerated, CBD can cause side effects, such as dry mouth, diarrhea, reduced appetite, drowsiness, and fatigue. CBD can also interact with other medications you are taking, such as blood thinners.

Another cause for concern is the unreliability of the purity and dosage of CBD in products. A recent study of 84 CBD products bought online showed that more than a quarter of the products contained less CBD than labeled. In addition, THC was found in 18 products. If you plan to use products containing CBD, talk to your primary health care provider.

People take cannabidiol by mouth for anxiety, bipolar disorder, a muscle disorder called dystonia, seizures, multiple sclerosis, Parkinson's disease, and schizophrenia.

Cannabidiol is possibly safe when taken by mouth and appropriately in adults. Cannabidiol doses of up to 300 mg daily have been used safely for up to 6 months. Higher doses of 1200-1500 mg daily have been used safely for up to 4 weeks. Cannabidiol sprays used under the tongue have been used in doses of 2.5 mg for up to 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years of age or older who can provide informed consent
2. Ability to read and write in the English language and follow study-related procedures
3. Ability to have mail/ study drug delivered to an address and/or P.O. Box in the recipient's name.
4. If a woman of childbearing age, willing to use a dual method of contraception (barrier and/or hormonal)

Exclusion Criteria:

1. Active illicit or non-prescribed drug use
2. Concomitant use of benzodiazepines
3. Concomitant use of Antabuse
4. Documented history and active treatment for seizure disorder
5. Transaminase elevation
6. Hepatitis C infection (currently on therapy and/or any transaminitis elevation)
7. Hepatitis B infection (currently on therapy and/or any transaminitis elevation)
8. Any form of mental impairment that will/could hinder safe participation in the study
9. Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety scores | 112 days (4-months)
  Generalized Anxiety Disorder (GAD-7), measure for anxiety. Baseline scores will be compared to scores at end of study across arms. Change in anxiety scores from baseline to end of study will be measured. Range from 0-4 for minimal; 5-9 mild; 10-14 moderate; 15-21 severe. Changes will be compared across arms. Increased scores will indicate that study product was not effective in decreasing symptoms measured (anxiety).
Depression scores | 112 days (4-months)
  Patient Health Questionnaire (PHQ-9), measure for depression. Change in depression scores from baseline to end of study.
  Total Score for Depression Severity will be compared across arms from baseline to end of study at 112-days.
  Score ranges from:
  1-4 Minimal depression; 5-9 Mild depression; 10-14 Moderate depression; 15-19 Moderately severe depression; 20-27 Severe depression. Increased scores indicate that study product is not effective in decreasing symptoms measured (depression).
Alcohol craving scores | 112 days (4-months)
  The Alcohol Craving Questionnaire Short Form (ACQ-SF-R) will be compared from baseline to end of study.
  Changes in craving score will be measured in each arm of study. Scores from 1-7 (strongly disagree to strongly agree) is measured across 12 items and 4 sub-scales ([1] compulsivity, [2] expectancy, [3] purposefulness, and [4] emotionality).
  The sum of the raw scores for each factor will be calculated and compared from baseline to the end of study across arms.
  Increased scores indicate that study product is not effective in reducing cravings for alcohol.

SECONDARY OUTCOMES:
To determine CBDs impact on anxiety, depression, and alcohol craving that trigger desires to consume alcohol versus abstain. | 112 days (4-months)
  Daily diary of symptom(s), dose(s) of study product and alcohol use will be kept by participants.
  Diary entries of symptoms, daily dose of study product and daily alcohol use will be measured and compared across study arms from baseline to end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P Young, PhD NP, Principal Investigator — Michael D Steward, MD + Thomas P Young, PhD, NP
Locations (1):
- Thomas P Young, PhD, NP, Novato, California, United States

IPD SHARING:
Plan to Share IPD: No
Not applicable/none planned

REFERENCES:
- [Result] Everitt BJ, Robbins TW. Neural systems of reinforcement for drug addiction: from actions to habits to compulsion. Nat Neurosci. 2005 Nov;8(11):1481-9. doi: 10.1038/nn1579. PMID 16251991
- [Result] Grotenhermen F. Pharmacokinetics and pharmacodynamics of cannabinoids. Clin Pharmacokinet. 2003;42(4):327-60. doi: 10.2165/00003088-200342040-00003. PMID 12648025
- [Result] MacCallum CA, Russo EB. Practical considerations in medical cannabis administration and dosing. Eur J Intern Med. 2018 Mar;49:12-19. doi: 10.1016/j.ejim.2018.01.004. Epub 2018 Jan 4. PMID 29307505
- [Result] Moreira FA, Lutz B. The endocannabinoid system: emotion, learning and addiction. Addict Biol. 2008 Jun;13(2):196-212. doi: 10.1111/j.1369-1600.2008.00104.x. Epub 2008 Apr 16. PMID 18422832
- [Result] Parsons LH, Hurd YL. Endocannabinoid signalling in reward and addiction. Nat Rev Neurosci. 2015 Oct;16(10):579-94. doi: 10.1038/nrn4004. Epub 2015 Sep 16. PMID 26373473
- [Result] Laviolette SR, Grace AA. The roles of cannabinoid and dopamine receptor systems in neural emotional learning circuits: implications for schizophrenia and addiction. Cell Mol Life Sci. 2006 Jul;63(14):1597-613. doi: 10.1007/s00018-006-6027-5. PMID 16699809
- See also: Background and summary of legislative Bill on HEMP production and cannabidiol (CBD) — https://www.fda.gov/news-events/congressional-testimony/hemp-production-and-2018-farm-bill-07252019
- See also: CannMed promotes understanding of cannabis' complex science and its medical benefits for patients in need. Since its founding, cannabis researchers & industry leaders collaborates with CannMed to announce their latest findings. — https://cannmedevents.com/